CLINICAL TRIAL: NCT01964703
Title: Effect of Rubus Occidentalis Extract on Plasma Glucose Levels in Subject With Prediabetes; A Proof-of-concept, Randomized, Double-blind, Parallel-group Placebo-controlled Study
Brief Title: Effect of Rubus Occidentalis Extract on Plasma Glucose Levels in Subject With Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sin Gon Kim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ED13024
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Prediabetes (Impaired Fasting Glucose and/or Impaired Glucose Tolerance)
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (Placebo Comparator)
- Rubus occidentalis extract 900mg (Active Comparator): taking Rubus occidentalis extract 900mg/day for 12weeks
  Interventions: Drug: Rubus occidentalis extract
- Rubus occidentalis extract 1800mg (Active Comparator): taking Rubus occidentalis extract 1800mg/day for 12weeks
  Interventions: Drug: Rubus occidentalis extract

INTERVENTIONS:
Drug: Rubus occidentalis extract
  Arms: Rubus occidentalis extract 1800mg; Rubus occidentalis extract 900mg

SUMMARY:
The purpose of this study is to determine whether Rubus occidentalis extract could improve fasting or postprandial serum glucose levels, and related metabolic markers among patients with prediabetes (impaired fasting glucose and/or impaired glucose tolerance).

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* prediabetes (fasting plasma glucose 100-125mg/dl, and/or post 75g OGTT plasma glucose 140-199mg/dl)

Exclusion Criteria:

* pregnant women
* taking anti-hyperglycemic agents within 3 months at the time of enrollment
* history of heart failure, myocardial infarction, cerebral infarction
* uncontrolled hypertension (systolic BP > 160mmHg, or diastolic BP > 100mmHg)
* serum triglyceride level > 500mg/dl
* kidney dysfunction (serum Creatinine > 30% of upper normal limits)
* hepatic dysfunction (AST, ALT > 3 times of upper normal limits)
* taking systemic glucocorticoids within 1 month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
serum glucose (fasting and post 75g oral glucose tolerance test) | 12 weeks

SECONDARY OUTCOMES:
serum insulin | 12 weeks

OTHER OUTCOMES:
HOMA IR, QUICKI, HOMA beta, lipid profile, inflammatory markers | 12 weeks

REFERENCES:
- [Derived] An JH, Kim DL, Lee TB, Kim KJ, Kim SH, Kim NH, Kim HY, Choi DS, Kim SG. Effect of Rubus Occidentalis Extract on Metabolic Parameters in Subjects with Prediabetes: A Proof-of-concept, Randomized, Double-blind, Placebo-controlled Clinical Trial. Phytother Res. 2016 Oct;30(10):1634-1640. doi: 10.1002/ptr.5664. Epub 2016 Jun 9. PMID 27279471